CLINICAL TRIAL: NCT00004659
Title: Phase II Randomized Study of Stereotactic Radiosurgery Plus Fractionated Whole-Brain Radiotherapy Vs Fractionated Whole-Brain Radiotherapy Alone for Multiple Primary or Metastatic Brain Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: University of Pittsburgh (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/11858; UPPUH-9511117
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-03

CONDITIONS: Brain Neoplasms
Keywords: adult brain tumor; brain tumor; childhood brain tumor; genetic condition; nervous tissue tumors; oncologic disorders; rare disease
MeSH Terms: conditions — Brain Neoplasms; Genetic Diseases, Inborn; Rare Diseases | interventions — Radiation; Radiosurgery

INTERVENTIONS:
Procedure: irradiation
Procedure: radiosurgery

SUMMARY:
OBJECTIVES: I. Evaluate whether stereotactic radiosurgery provides local control at multiple sites in patients with primary or metastatic brain tumors, controlled systemic disease, and preserved neurologic function.

II. Examine survival, clinical outcome, and local tumor imaging response in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Tumor size and number are confirmed prior to randomization. Patients are stratified by participating institution.

Patients are randomly assigned to 1 of 2 treatment groups. One group is treated with fractionated whole-brain irradiation using megavoltage equipment.

The second group receives stereotactic radiosurgery plus fractionated whole-brain radiotherapy. Stereotactic radiosurgery involves irradiation of all tumors to the margins on stereotactic computerized tomography or magnetic resonance imaging. Either treatment may be administered first; the second treatment begins within 1 month of the first.

Concurrent anticonvulsants and steroids are allowed. Patients are followed for change in size and number of tumors at 1, 3, and 6 months; follow-up clinical exams are performed at least every 2 months.

ELIGIBILITY:
* Multiple newly diagnosed brain tumors
* Histologic confirmation of carcinoma at primary or metastatic site
* Tumors less than 25 mm mean diameter and more than 5 mm from optic chiasm
* No more than 4 tumors on magnetic resonance imaging
* Systemic disease controlled
* Neurologic function preserved
* Radiographic staging within 2 months of randomization required
* Performance status: Karnofsky 70%-100%

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 1994-11

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Kondziolka, Study Chair — University of Pittsburgh